CLINICAL TRIAL: NCT04079660
Title: Prospective, Observational Study Evaluating the Glycemic Control Based on Serum Fructosamine Concentration vs. hemoglobinA1c (HbA1c) in Diabetic Patients Undergoing Surgeries
Brief Title: Glycemic Control Based on Serum Fructosamine Concentration vs. hemoglobinA1c (HbA1c) in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Barbara Rogers, Associate Professor, Ohio State University
Other Study IDs: 2018H0320
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Diabetes
Keywords: hemoglobinA1c; serum fructosamine; glycemic control
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical patients: Diabetic patients scheduled to undergo non-cardiac surgery
  Interventions: Diagnostic Test: Capillary blood glucose blood draw

INTERVENTIONS:
Diagnostic Test: Capillary blood glucose blood draw — Capillary blood glucose (CBG), HbA1c, fructosamine, albumin, BUN, and creatinine values will be obtained from a blood draw as a standard of care
  Other Names: CBG

SUMMARY:
Diabetes mellitus is associated with negative outcomes in patients undergoing surgery. Blood sugar levels are monitored by measuring a values that include but are not limited to hemoglobin A1c, capillary blood glucose, and fructosamine . This study is being done to investigate if there is an associated between these values and postsurgical outcomes.

DETAILED DESCRIPTION:
This study aims to compare the predictive capacity of both fructosamine and HbA1c on preoperative basal glucose level, as well as adverse events (cardiovascular events, surgical site infection, and mortality) and length of post-anesthesia care unit (PACU) stay in both Type I and Type II diabetic patients. Secondary outcomes include length of anesthesia administration, an indicator of intraoperative complications, and perioperative glucose level.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients able to consent.
2. Patients with either Type I or Type II diabetes mellitus (DM)
3. Patients undergoing non-cardiac surgeries under general anesthesia
4. ≥ 18 years of age

Exclusion Criteria:

1. Inability to read, understand or sign the consent form
2. End-stage renal disease
3. Special populations (Incarcerated individuals, pregnant female patients)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Diabetic patients sover 18 years of age, scheduled to undergo surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
fasting capillary blood glucose level | 1 hour
  Association between pre-operative HbA1c and fructosamine with pre-operative, fasting capillary blood glucose level measured the morning of surgery in preoperative holding area.

SECONDARY OUTCOMES:
hypoglycemia | 1 day
  i. Incidence of hypoglycemia, defined as CBG < 70 mg/dL, during the perioperative period
hyperglycemia | 1 day
  ii. Incidence of hyperglycemia, defined as CBG > 180 mg/dL, during the perioperative period
infection | 1 day
  Incidence of wound infection
wound healing | 1 day
  Incidence of poor wound healing
delirium | 1 day
  Incidence of post-operative delirium
reoperation | 1 day
  Incidence of reoperation procedure
LOS | 1 day
  Length of PACU stay

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Background] Miller JD, Richman DC. Preoperative Evaluation of Patients with Diabetes Mellitus. Anesthesiol Clin. 2016 Mar;34(1):155-69. doi: 10.1016/j.anclin.2015.10.008. PMID 26927745
- [Background] Frisch A, Chandra P, Smiley D, Peng L, Rizzo M, Gatcliffe C, Hudson M, Mendoza J, Johnson R, Lin E, Umpierrez GE. Prevalence and clinical outcome of hyperglycemia in the perioperative period in noncardiac surgery. Diabetes Care. 2010 Aug;33(8):1783-8. doi: 10.2337/dc10-0304. Epub 2010 Apr 30. PMID 20435798
- [Background] Shohat N, Tarabichi M, Tischler EH, Jabbour S, Parvizi J. Serum Fructosamine: A Simple and Inexpensive Test for Assessing Preoperative Glycemic Control. J Bone Joint Surg Am. 2017 Nov 15;99(22):1900-1907. doi: 10.2106/JBJS.17.00075. PMID 29135663
- [Background] van den Boom W, Schroeder RA, Manning MW, Setji TL, Fiestan GO, Dunson DB. Effect of A1C and Glucose on Postoperative Mortality in Noncardiac and Cardiac Surgeries. Diabetes Care. 2018 Apr;41(4):782-788. doi: 10.2337/dc17-2232. Epub 2018 Feb 13. PMID 29440113
- [Background] Maradit Kremers H, Lewallen LW, Mabry TM, Berry DJ, Berbari EF, Osmon DR. Diabetes mellitus, hyperglycemia, hemoglobin A1C and the risk of prosthetic joint infections in total hip and knee arthroplasty. J Arthroplasty. 2015 Mar;30(3):439-43. doi: 10.1016/j.arth.2014.10.009. Epub 2014 Oct 15. PMID 25458090
- [Background] Danese E, Montagnana M, Nouvenne A, Lippi G. Advantages and pitfalls of fructosamine and glycated albumin in the diagnosis and treatment of diabetes. J Diabetes Sci Technol. 2015 Mar;9(2):169-76. doi: 10.1177/1932296814567227. Epub 2015 Jan 14. PMID 25591856
- [Background] Kowalczuk-Wieteska AM, Wrobel M, Rokicka D, Szymborska-Kajanek A, Foremny J, Nadziakiewicz P, Zembala M, Strojek K. Determination of the value of glycated hemoglobin HbA1c and fructosamine in assessing the risk of perioperative complications after cardiac surgery in patients with type 2 diabetes. Kardiochir Torakochirurgia Pol. 2016 Dec;13(4):305-308. doi: 10.5114/kitp.2016.64869. Epub 2016 Dec 30. PMID 28096825
- [Background] Malmstrom H, Walldius G, Grill V, Jungner I, Gudbjornsdottir S, Hammar N. Fructosamine is a useful indicator of hyperglycaemia and glucose control in clinical and epidemiological studies--cross-sectional and longitudinal experience from the AMORIS cohort. PLoS One. 2014 Oct 29;9(10):e111463. doi: 10.1371/journal.pone.0111463. eCollection 2014. PMID 25353659
- [Background] Rodriguez-Segade S, Rodriguez J, Camina F. Corrected Fructosamine improves both correlation with HbA1C and diagnostic performance. Clin Biochem. 2017 Feb;50(3):110-115. doi: 10.1016/j.clinbiochem.2016.10.014. Epub 2016 Oct 21. PMID 27777100
- [Background] Constanti C, Simo JM, Joven J, Camps J. Serum fructosamine concentration in patients with nephrotic syndrome and with cirrhosis of the liver: the influence of hypoalbuminaemia and hypergammaglobulinaemia. Ann Clin Biochem. 1992 Jul;29 ( Pt 4):437-42. doi: 10.1177/000456329202900412. PMID 1642452
- [Background] Gan T, Liu X, Xu G. Glycated Albumin Versus HbA1c in the Evaluation of Glycemic Control in Patients With Diabetes and CKD. Kidney Int Rep. 2017 Nov 21;3(3):542-554. doi: 10.1016/j.ekir.2017.11.009. eCollection 2018 May. PMID 29854962
- [Background] American Diabetes Association. 6. Glycemic Targets: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018 Jan;41(Suppl 1):S55-S64. doi: 10.2337/dc18-S006. PMID 29222377